CLINICAL TRIAL: NCT01585051
Title: Effect of Administration of 25(OH) Vitamin on Mean 24 Hour Blood Pressure and HBA1c Levels in Patients With Stable Type 2 Diabetes Mellitus
Brief Title: Effect of Vitamin D Supplementation on Blood Pressure and HbA1c Levels in Patients With T2D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Principal Investigator, Reto Krapf, Professor of Medicine, Kantonsspital Baselland Bruderholz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: x335/08
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus Type 2
Keywords: vitamin D; blood pressure; typ 2 diabetes mellitus; blood glucose; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vitamin D; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Active Comparator): Intervention: Intramuscular injection of 300 000 U of 25(OH)vitamin D
  Interventions: Drug: 25(OH) vitamin D
- placebo (Placebo Comparator): administration of 0.9 % NaCl as a placebo
  Interventions: Drug: 0.9 % NaCl

INTERVENTIONS:
Drug: 25(OH) vitamin D — 300 000 U intramuscularly, one dosage, in subjects with 25 (OH) vit D levels below 80 nmol/L, another dosage of 150 000 U after 3 months if 25(OH)vit D levels continue to be below 80 nmol/L.
  Arms: vitamin D
Drug: 0.9 % NaCl — 1 ml of 0.9 % of NaCl at the beginning and 0.5 ml of 0.9 % NaCl after three months
  Arms: placebo

SUMMARY:
The effect of administration of vitamin D is tested on the long-term control of blood sugar (as measured by HbA1-c levels in blood) and mean blood pressure (as measured by 24 hour blood pressure profiles)in patients with stable type 2 diabetes mellitus

ELIGIBILITY:
Inclusion criteria

* Men and women, ages ≥18 years
* Official diagnostic criteria for type 2 diabetes fulfilled in patients on any type of oral or parenteral glucose-lowering treatment
* Independent living at home
* On stable regimen of BP meds (if any) with BP well controlled and/or K supplement (if any) for 2 months and which is deemed unlikely to change during the study
* Stable glucose control for 2 months by any approved method including insulin

Exclusion criteria

* Patients with type 1 diabetes (or insulin-requiring diabetes of unclear type)
* Patients on hemodialysis, with hyperparathyroidism or active cancer disease
* Patients with known metabolic bone disease
* Laboratory evidence of kidney (eGFR < 60 ml/min) or liver disease
* Dietary calcium intake exceeding 1500mg/d (as estimated by dietary history)
* 25(OH) vitamin D levels at baseline > 70 nmol/L
* Calciuria (> 8 mmol/24 hours as measured by 24 hour urine collections)
* Hypo- and hypercalcemias and hypo- and hyperphosphatemias of any cause
* Medications that affect vitamin D metabolism (e.g. antiepileptic drugs, calcimimetics, 1-34 PTH (Forsteo) vitamin D therapy over and above 400U daily 6 months prior to enrollment and during the study)
* Foreseeable need for adaptation of either glucose- or blood pressure lowering during the next 6 months as decided by the family physician or the treating diabetologist - see above
* History of binge eating or wt gain or loss exceeding 6 kg in past 18 months
* Patients on any type of inhibitors of plasma coagulation (i.e. coumarine, heparins)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in HBA1-c levels | 3 and 6 months
24 hour mean blood pressure | 3 and 6 months

SECONDARY OUTCOMES:
plasma glucose | 3 and 6 months
HOMA | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Reto Krapf, MD, Principal Investigator — Department of Medicine, Kantonsspital Bruderholz, University of Basel, Switzerland
Locations (1):
- Department of medicine, Kantonsspital Bruderholz, Bruderholz/Basel, Basel-Landschaft, Switzerland

REFERENCES:
- [Derived] Jehle S, Lardi A, Felix B, Hulter HN, Stettler C, Krapf R. Effect of large doses of parenteral vitamin D on glycaemic control and calcium/phosphate metabolism in patients with stable type 2 diabetes mellitus: a randomised, placebo-controlled, prospective pilot study. Swiss Med Wkly. 2014 Mar 20;144:w13942. doi: 10.4414/smw.2014.13942. PMID 24652692